CLINICAL TRIAL: NCT02178046
Title: Non-Invasive Oral Biofilm Characterization
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Petra Wilder-Smith, DDS., PhD., Professor, Director of Dentistry, University of California, Irvine
Other Study IDs: 20141167
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Gingivitis
Keywords: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gingivitis: optical measurements
  Interventions: Device: optical measurements

INTERVENTIONS:
Device: optical measurements — Laser Speckle Imaging, Optical Coherence Tomography and Multiphoton Microscopy

SUMMARY:
There is a need for toothpastes that more effectively remove oral plaque and prevent re-formation. The objective of this study is to map the development and resolution of clinical gingivitis using conventional clinical examination and imaging data to determine how useful imaging techniques can be for evaluating how well a toothpaste cleans the teeth

DETAILED DESCRIPTION:
The researcher can use imaging techniques to map changes in gingival blood flow during the development and resolution of fully reversible, early clinical gingivitis using standard-of-care clinical indices as gold standard

The researcher can use imaging techniques to map inflammatory microstructural changes in the oral mucosa including swelling, vasodilation and edema during the development and resolution of fully reversible, early clinical gingivitis using standard-of-care clinical indices as gold standard

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female 18-25 years of age
* Volunteers with gingivitis but no periodontitis

Exclusion Criteria:

* Subjects who must receive dental treatment during the study dates.
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouth rinses. Allergy to personal care/consumer products or their ingredients.
* Individuals who have taken antibiotics in the previous 3 months
* Individuals who are pregnant or nursing

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population will be selected from UCI Medical Center a referral base for dentists in the greater Orange County area for diagnosis of patients with suspected intra-oral lesions. The UCI student dental health clinic caters to UCI students, staff and faculty.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Changes in gingival perfusion | up to 6 weeks
  optical measurements

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wilder-Smith, DDS. PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute, Irvine, California, United States